CLINICAL TRIAL: NCT07238868
Title: A Multicenter, Open-label, Long-term, Safety, Tolerability, and Efficacy Study of CB03-154 in Subjects Diagnosed With Epilepsy
Brief Title: An Open-label Study to Evaluate Safety, Tolerability, and Efficacy of CB03-154 in Subjects Diagnosed With Epilepsy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB03-154-EP202
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Subjects from CB03-154-EP201 (Experimental): The subjects who completed the CB03-154-EP201 will be enrolled and begin with a two-week course of CB03-154 at 10 mg QD. Upon demonstrating good tolerability, the dose will be increased to 20 mg QD and continued for up to two years.
  Interventions: Drug: CB03-154

INTERVENTIONS:
Drug: CB03-154 — All enrolled subjects will begin with a two-week course of CB03-154 at 10 mg QD. Upon demonstrating good tolerability, the dose will be increased to 20 mg QD and continued for up to two years.

SUMMARY:
CB03-154 is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Focal Epilepsy.

DETAILED DESCRIPTION:
This is an open-label extension study based on the Phase 2 clinical trial CB03-154-EP201. The study aims to assess the long-term safety, tolerability, efficacy, and pharmacokinetics (PK) of CB03-154 at a maximum dose of 20 mg administered orally once daily (QD) in patients with epilepsy. Eligible subjects are those who successfully completed the prior CB03-154-EP201 study without early discontinuation. The treatment in this extension study will last for up to two years.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject must be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study.

  2. Subject must have successfully completed the DBP and have not terminated early from Study CB03-154-EP201, met all eligibility requirements, and had no important protocol deviations (in the opinion of the sponsor) or AEs (in the opinion of the investigator) that would preclude the subject's entry into the long-term extension study, and judged to be efficacious based on the blinded data review (in the opinion of the investigator).

  3. In the opinion of the investigator, the subject is able to understand verbal and written instructions and will adhere to all study schedules and requirements.

  4. Subject is able to keep accurate seizure diaries.

Exclusion Criteria:

- 1. Subject met any of the withdrawal criteria while in Study CB03-154-EP201. 2. Subject has any medical condition, personal circumstance, or ongoing AE (from Study CB03-154-EP201) that, in the opinion of the investigator, exposes the subject to unacceptable risk by participating in the study, or prevents adherence to the protocol.

3. Subject is planning to enter a clinical study with a different investigational drug or planning to use any experimental device for treatment of epilepsy during the study and until 28 days after completion of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
To assess the long-term tolerability and safety of CB03-154 in patients diagnosed with epilepsy. | In the entire period of the whole study, including a treatment period up to 2 years (104 weeks) and a post treatment follow-up period of 8 weeks.
  Severity and frequency of associated AEs/serious adverse events (SAEs)
To assess the long-term efficacy of CB03-154 in patients diagnosed with epilepsy. | In the entire period of the whole study, including a treatment period up to 2 years (104 weeks) and a post treatment follow-up period of 8 weeks.
  Median percent change (MPC) in monthly (28 days) seizure frequency from baseline (the end of the DBP of study CB03 154-EP201) to the entire treatment period.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax). | In the Week 2±3 days , Week 4±3 days , Week 13±3 days , and Week 26±7 days.
  For all subjects, blood samples will be obtained at Week 2, Week 4, Week 13, and Week 26 for in the period of study for plasma concentration measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No